CLINICAL TRIAL: NCT00607295
Title: Prospective Randomized Study on Efficacy and Safety of Clino-san® in the Management of Vaginal Dryness in Breast Cancer Patients
Brief Title: Efficacy and Safety of Clino-san on Vaginal Dryness of Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Yookyung Lee, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SNUH-OG-07-211
Record Dates: First submitted 2008-02-04; First posted 2008-02-05 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer; Vaginal Atrophy
Keywords: chemotherapy; hormonal therapy; urogenital atrophy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Clino-san 2ml vaginal application 3 times per week for 12 weeks
  Interventions: Drug: clino-san vaginal lubricant
- 2 (Placebo Comparator): placebo 2ml vaginal application 3 times per week for 12 weeks
  Interventions: Drug: clino-san vaginal lubricant

INTERVENTIONS:
Drug: clino-san vaginal lubricant — Clino-san 2ml vaginal application 3 times per week for 12 weeks

SUMMARY:
1. Although after treatment for breast cancer such as chemotherapy or hormonal therapy, urogenital atrophy is common, the patients are seldomly treated for several reasons. Management of this problem is important for improving quality of life.
2. "Clino-san" is a kind of vaginal lubricant with pH 5 which is similar pH of premenopausal vaginal discharge. After randomization of patients, they are treated with Clino-san or placebo 3 times/week for 12 weeks.
3. We check the vaginal symptoms, vag dryness severity score, and ultrasonography at baseline, 4, 8, and 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients
* who are treated with chemotherapy or hormonal therapy
* who experience no menstruation after the previous therapy
* who complain of vaginal dryness

Exclusion Criteria:

* other cancer patients
* other severe disease
* poor compliance

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
vaginal dryness score | for 12 weeks

SECONDARY OUTCOMES:
sexual dysfunction | for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jae Weon Kim, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee YK, Chung HH, Kim JW, Park NH, Song YS, Kang SB. Vaginal pH-balanced gel for the control of atrophic vaginitis among breast cancer survivors: a randomized controlled trial. Obstet Gynecol. 2011 Apr;117(4):922-927. doi: 10.1097/AOG.0b013e3182118790. PMID 21422866